CLINICAL TRIAL: NCT03228264
Title: A Randomized Controlled, Evaluator-blinded, Multi-center Trial Investigating Telerehabilitation as an add-on to Face-to-face Speech and Language Therapy in Post-stroke Aphasia.
Brief Title: A Trial Investigating Telerehabilitation as an add-on to Face-to-face Speech and Language Therapy in Post-stroke Aphasia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-01577
Record Dates: First submitted 2017-07-12; First posted 2017-07-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Aphasia; Chronic Stroke; Post Stroke Seizure
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized, controlled, evaluator-blinded multi-center superiority trial with two parallel groups and with word finding ability as primary endpoint at the end of the intervention. Aphasia outpatients will be recruited and randomly assigned to the experimental or control group. The randomization will be stratified by the study centre (Bern, Luzern) and the severity of aphasia (mild with a raw value/T-value smaller than 5/52, severe with a raw value/T-value greater or equal to 5/52 for the Token Test). Both groups will do a four weeks intensive tablet-delivered telerehabilitation training (2 hours a day).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High teleSLT frequency (Experimental): During four weeks all patients will do a daily two-hour training session with a tablet computer (consisting of teleSLT and teleCT) at their home. In the experimental group 80% of the training time will be devoted to teleSLT and 20% to teleCT. Both groups receive the same amount of ucSLT.
  Interventions: Device: teleSLT; Device: teleCT
- Low teleSLT frequency (Active Comparator): During four weeks all patients will do a daily two-hour training session with a tablet computer (consisting of teleSLT and teleCT) at their home. In the control group 20% of the training time will be devoted to teleSLT and 80% to teleCT. Both groups receive the same amount of ucSLT.
  Interventions: Device: teleSLT; Device: teleCT

INTERVENTIONS:
Device: teleSLT — The teleSLT intervention consists of a daily training session with a tablet computer at the patients' home. The teleSLT application that will be used for this study was developed within a multidisciplinary team of speech and language therapists, neurologists and computer engineers that have transferred well-established SLT exercises to a tablet computer. The investigators call this application Bern Aphasia App (BAA). During the four weeks the training time with the BAA differs between the two arms. The experimental group trains for 96 minutes per day (80% of two hours) and the control group for 24 minutes per day (20% of two hours).
Device: teleCT — For the cognitive training the investigators will use two custom-made versions of popular commercial casual puzzle video games: Flow Free (Big Duck Games LCC) and Bejeweled (PopCap Games). The video games are also delivered on tablet-computers. Again, during the four weeks the training time differs between the two arms. The experimental group trains for 24 minutes and the control group for 96 minutes per day.

SUMMARY:
The aim of this study is to investigate the effects of high-frequency short duration tablet-based speech and language therapy (teleSLT) mixed with cognitive training (teleCT) in chronic stroke patients. Recent studies suggest that chronic stroke patients benefit from SLT with high frequency and that cognitive abilities can play a role in sentence comprehension and production by individuals with aphasia. To investigate the effects of the distribution of training time for teleSLT and teleCT the investigators use two combinations. In the experimental group 80% of the training time will be devoted to teleSLT and 20% to teleCT whereas in the control group 20% of the training time will be devoted to teleSLT and 80% to teleCT. Both groups receive the same total amount and frequency of intervention but with different distributions. At three time points (pre-, post-test and 8 week follow-up) the patients' word finding ability is measured.

DETAILED DESCRIPTION:
A recent Cochrane intervention review revealed evidence for the effectiveness of using speech and language therapy (SLT) for people with aphasia following stroke in terms of functional communication, receptive and expressive language. The authors highlight positive effects of higher training frequency on functional outcome. Also other authors emphasizes the importance of training frequency. In the meta-analysis with 968 patients the authors found that only intervention studies with more than five hours training per week lead to positive effects on speech and language function. They highlighted that it might be better to train short but with a high frequency than long with a low frequency. While some researchers emphasizes the benefit of early intervention, several studies found that also chronic stroke patients can benefit from intensive SLT. One possible approach to increase training frequency and duration is to complement therapist delivered usual care SLT (ucSLT) with telerehabilitation SLT (teleSLT) delivered in the patient's home.

Aphasia is frequently accompanied by deficits of working memory (WM), speed of processing (SP) and executive functions (EF). Recent studies suggest that these cognitive abilities can play a role in sentence comprehension and production by individuals with aphasia and that WM, SP and EF can be enhanced with intensive practice. The authors suggest that SLT therapy should be accompanied with cognitive training (CT). It remains however unclear what percentage of the training time should be devoted to SLT and to cognitive training respectively. For the current study the investigators will use two combinations of teleSLT and telerehabilitation cognitive training (teleCT), where one combination will have a higher percentage of time devoted to teleSLT and the other a higher percentage devoted to teleCT. The latter will serve as the control group to examine the effect of teleSLT.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over.
* Diagnosis of stroke, onset of stroke at least 3 months prior to inclusion
* Diagnosis of aphasia due to stroke, as confirmed by a speech and language therapist.
* Raw value for the German version of the Token Test (De Renzi & Vignolo, 1962) has to be smaller or equal to 8 (T-value smaller or equal to 60).
* Sufficient vision and cognitive ability to work with the teleSLT software (a simple matching task on the tablet computer will be used to test this).
* Written informed consent.

Exclusion Criteria:

* Any other pre-morbid speech and language disorder caused by a deficit other than stroke.
* Requirement for treatment in language other than German.
* Currently using a computer speech therapy software.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Understandability of verbal communication | Pre-test (Baseline, week 0)
  The understandability of verbal communication is assessed with the A-scale of the Amsterdam-Nijmegen Everyday Language Test (ANELT). For this scale, oral answers in ten everyday life scenarios are scored with respect to understandability of the message, i.e. the content of the message independent of the linguistic form of the utterance (Blomert, Kean, Koster, & Schokker, 1994). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the beginning of the intervention.
Understandability of verbal communication | Post-test (Change from Baseline at week 4)
  The understandability of verbal communication is assessed with the A-scale of the Amsterdam-Nijmegen Everyday Language Test (ANELT). For this scale, oral answers in ten everyday life scenarios are scored with respect to understandability of the message, i.e. the content of the message independent of the linguistic form of the utterance (Blomert, Kean, Koster, & Schokker, 1994). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the end of the intervention.
Understandability of verbal communication | 8 week follow-up (Change from Baseline at week 12)
  The understandability of verbal communication is assessed with the A-scale of the Amsterdam-Nijmegen Everyday Language Test (ANELT). For this scale, oral answers in ten everyday life scenarios are scored with respect to understandability of the message, i.e. the content of the message independent of the linguistic form of the utterance (Blomert, Kean, Koster, & Schokker, 1994). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place eight weeks after the intervention.

SECONDARY OUTCOMES:
Intelligibility of verbal communication | Pre-test (Baseline, week 0)
  The intelligibility of verbal communication is assessed with the B-scale of the Amsterdam-Nijmegen Everyday Language Test (ANELT). For this scale, oral answers in ten everyday life scenarios (same situation as for the A-scale of ANELT) are scored with respect to the intelligibility of the utterance, i.e. the perception of the utterance independent of the content or the meaning (Blomert et al., 1994). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the beginning of the intervention.
Intelligibility of verbal communication | Post-test (Change from Baseline at week 4)
  The intelligibility of verbal communication is assessed with the B-scale of the Amsterdam-Nijmegen Everyday Language Test (ANELT). For this scale, oral answers in ten everyday life scenarios (same situation as for the A-scale of ANELT) are scored with respect to the intelligibility of the utterance, i.e. the perception of the utterance independent of the content or the meaning (Blomert et al., 1994). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the end of the intervention.
Intelligibility of verbal communication | 8 week follow-up (Change from Baseline at week 12)
  The intelligibility of verbal communication is assessed with the B-scale of the Amsterdam-Nijmegen Everyday Language Test (ANELT). For this scale, oral answers in ten everyday life scenarios (same situation as for the A-scale of ANELT) are scored with respect to the intelligibility of the utterance, i.e. the perception of the utterance independent of the content or the meaning (Blomert et al., 1994). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place eight weeks after the intervention.
Impairment specific language measures | Pre-test (Baseline, week 0)
  The impairment specific language measures are assessed with "Sprachsystematisches APhasie Screening" (SAPS). The SAPS assesses comprehension (receptive) and production (expressive) abilities in the domains of phonetics and phonology (sub-lexical level), lexicon and semantic (lexical level) and morphology and syntax (morpho-syntactic level). For both modules (receptive and expressive) all three levels are divided into three difficulty levels. Based on these assessed comprehension and production abilities on all three levels it is possible to derive and evaluate disorder specific treatments (Blömer, Pesch, Willmes, Huber, Springer, & Abel, 2013). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the beginning of the intervention.
Impairment specific language measures | Post-test (Change from Baseline at week 4)
  The impairment specific language measures are assessed with "Sprachsystematisches APhasie Screening" (SAPS). The SAPS assesses comprehension (receptive) and production (expressive) abilities in the domains of phonetics and phonology (sub-lexical level), lexicon and semantic (lexical level) and morphology and syntax (morpho-syntactic level). For both modules (receptive and expressive) all three levels are divided into three difficulty levels. Based on these assessed comprehension and production abilities on all three levels it is possible to derive and evaluate disorder specific treatments (Blömer, Pesch, Willmes, Huber, Springer, & Abel, 2013). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the end of the intervention.
Impairment specific language measures | 8 week follow-up (Change from Baseline at week 12)
  The impairment specific language measures are assessed with "Sprachsystematisches APhasie Screening" (SAPS). The SAPS assesses comprehension (receptive) and production (expressive) abilities in the domains of phonetics and phonology (sub-lexical level), lexicon and semantic (lexical level) and morphology and syntax (morpho-syntactic level). For both modules (receptive and expressive) all three levels are divided into three difficulty levels. Based on these assessed comprehension and production abilities on all three levels it is possible to derive and evaluate disorder specific treatments (Blömer, Pesch, Willmes, Huber, Springer, & Abel, 2013). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place eight weeks after the intervention.
Perceived quality of life | Pre-test (Baseline, week 0)
  The perceived quality of life is assessed with the Stroke and Aphasia Quality of Life Scale with 39 items in total (SAQOL-39) which is an interview-administered self-report scale consisting of the four subdomains physical, psychosocial, communication and energy (Hilari, Byng, & Smith, 2003). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the beginning of the intervention.
Perceived quality of life | Post-test (Change from Baseline at week 4)
  The perceived quality of life is assessed with the Stroke and Aphasia Quality of Life Scale with 39 items in total (SAQOL-39) which is an interview-administered self-report scale consisting of the four subdomains physical, psychosocial, communication and energy (Hilari, Byng, & Smith, 2003). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place at the end of the intervention.
Perceived quality of life | 8 week follow-up (Change from Baseline at week 12)
  The perceived quality of life is assessed with the Stroke and Aphasia Quality of Life Scale with 39 items in total (SAQOL-39) which is an interview-administered self-report scale consisting of the four subdomains physical, psychosocial, communication and energy (Hilari, Byng, & Smith, 2003). The measurement is performed in a face-to-face interaction between the patients and the evaluator and takes place eight weeks after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Nef, Prof. Dr., Principal Investigator — Gerontechnology and Rehabilitation, ARTORG Centre for Biomedical Engineering Research
Locations (2):
- Switzerland (2):
  - ARTORG Center for Biomedical Engineering Research, Bern
  - Center for Neurology and Neurorehabilitation, Lucerne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhogal SK, Teasell R, Speechley M. Intensity of aphasia therapy, impact on recovery. Stroke. 2003 Apr;34(4):987-93. doi: 10.1161/01.STR.0000062343.64383.D0. Epub 2003 Mar 20. PMID 12649521
- [Background] Brady MC, Kelly H, Godwin J, Enderby P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2012 May 16;(5):CD000425. doi: 10.1002/14651858.CD000425.pub3. PMID 22592672
- [Background] Caplan D, Waters G. Memory mechanisms supporting syntactic comprehension. Psychon Bull Rev. 2013 Apr;20(2):243-68. doi: 10.3758/s13423-012-0369-9. PMID 23319178
- [Background] Crotty M, George S. Retraining visual processing skills to improve driving ability after stroke. Arch Phys Med Rehabil. 2009 Dec;90(12):2096-102. doi: 10.1016/j.apmr.2009.08.143. PMID 19969174
- [Background] Kendall DL, Oelke M, Brookshire CE, Nadeau SE. The Influence of Phonomotor Treatment on Word Retrieval Abilities in 26 Individuals With Chronic Aphasia: An Open Trial. J Speech Lang Hear Res. 2015 Jun;58(3):798-812. doi: 10.1044/2015_JSLHR-L-14-0131. PMID 25766309
- [Background] Sandberg CW, Bohland JW, Kiran S. Changes in functional connectivity related to direct training and generalization effects of a word finding treatment in chronic aphasia. Brain Lang. 2015 Nov;150:103-16. doi: 10.1016/j.bandl.2015.09.002. Epub 2015 Sep 20. PMID 26398158
- [Background] Wang CP, Hsieh CY, Tsai PY, Wang CT, Lin FG, Chan RC. Efficacy of synchronous verbal training during repetitive transcranial magnetic stimulation in patients with chronic aphasia. Stroke. 2014 Dec;45(12):3656-62. doi: 10.1161/STROKEAHA.114.007058. Epub 2014 Nov 6. PMID 25378426
- [Background] Zakarias L, Keresztes A, Marton K, Wartenburger I. Positive effects of a computerised working memory and executive function training on sentence comprehension in aphasia. Neuropsychol Rehabil. 2018 Apr;28(3):369-386. doi: 10.1080/09602011.2016.1159579. Epub 2016 Mar 21. PMID 26999324
- [Background] Blomert L, Kean ML, Koster C, Schokker, J. Amsterdam-Nijmegen everyday language test: construction, reliability and validity. Aphasiology 8(4): 381-407, 1994.
- [Background] Blömer F, Pesch A, Willmes K, Huber W, Springer L, Abel S. Das sprachsystematische Aphasiescreening (SAPS): Konstruktionseigenschaften und erste Evaluierung. Zeitschrift für Neuropsychologie 24(3): 139-148, 2013.
- [Background] Hilari K, Byng S, Lamping DL, Smith SC. Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39): evaluation of acceptability, reliability, and validity. Stroke. 2003 Aug;34(8):1944-50. doi: 10.1161/01.STR.0000081987.46660.ED. Epub 2003 Jul 10. PMID 12855827
- [Background] DE RENZI E, VIGNOLO LA. The token test: A sensitive test to detect receptive disturbances in aphasics. Brain. 1962 Dec;85:665-78. doi: 10.1093/brain/85.4.665. No abstract available. PMID 14026018
- [Derived] Uslu AS, Gerber SM, Schmidt N, Rothlisberger C, Wyss P, Vanbellingen T, Schaller S, Wyss C, Koenig-Bruhin M, Berger T, Nyffeler T, Muri R, Nef T, Urwyler P. Investigating a new tablet-based telerehabilitation app in patients with aphasia: a randomised, controlled, evaluator-blinded, multicentre trial protocol. BMJ Open. 2020 Nov 11;10(11):e037702. doi: 10.1136/bmjopen-2020-037702. PMID 33177134